CLINICAL TRIAL: NCT02293447
Title: Intra-arterial Lidocaine for Pain Control Post Uterine Fibroid Embolization : a Single-center Prospective Randomized Study
Brief Title: Intra-arterial Lidocaine for Pain Control Post Uterine Fibroid Embolization
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Dheeraj Rajan, Attending Interventional Radiologist and Associate Professor, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 14-8053
Record Dates: First submitted 2014-11-10; First posted 2014-11-18 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Uterine Leiomyomas
Keywords: Uterine; Fibroid; Embolization; Leiomyoma; Lidocaine; Pain
MeSH Terms: conditions — Myofibroma; Leiomyoma; Pain | interventions — Anesthetics, Local; Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): The control group will undergo uterine artery embolization according to regular protocol, without the administration of lidocaine.
- Lidocaine per-embolization (Experimental): This group will receive 10mL of 1% lidocaine in both uterine artery during the embolization; the lidocaine will be mixed with the embolization particles.
  Interventions: Drug: Lidocaine per-embolization
- Lidocaine post-embolization (Experimental): 10mL of 1% lidocaine will be injected in both uterine arteries after embolization endpoint is achieved.
  Interventions: Drug: Lidocaine post-embolization

INTERVENTIONS:
Drug: Lidocaine per-embolization — 10mL of 1% lidocaine will be mixed with the embolization particles. Lidocaine will therefore be injected during the embolization.
  Other Names: Local anesthetic; Amide-type anesthetic; Lidocaine hydrochloride; 00884154
  Arms: Lidocaine per-embolization
Drug: Lidocaine post-embolization — 10mL of 1% lidocaine will be injected in both uterine arteries after the embolization endpoint is achieved.
  Other Names: Local anesthetic; Amide-type anesthetic; Lidocaine hydrochloride; 00884154
  Arms: Lidocaine post-embolization

SUMMARY:
Uterine artery embolization (UAE) is a minimally invasive treatment for women with symptomatic fibroids. It is similar to hysterectomy in term of satisfaction and symptoms improvement, with fewer complications and at lower cost. However, the majority of women undergoing UFE experience important pain after the procedure despite optimal analgesia, with one third reporting pain equal or worse than labor. Pain is the more common cause of prolonged hospital stay or readmission. There is need for a simple, efficient way to reduce post-procedural pain.

For this prospective randomized study, the hypothesis is that an anesthetic drug, lidocaine, injected in the uterine arteries diminishes pain post-UFE. Patients will be randomized in 3 groups: control, lidocaine injected during embolization, and lidocaine injected after embolization. Pain will be evaluated using a validated scale at 4h and 24h post-intervention. Hospital length-of-stay and total narcotic dose administered will be evaluated in the three groups.

This is the first Canadian study evaluating lidocaine use for pain control in UFE patients. Results will be transferable to clinical practice, considering the use of lidocaine is simple and cost is negligible. It could have a great impact on pain management in women undergoing UFE in all practice settings.

ELIGIBILITY:
Inclusion Criteria:

* Indication for uterine fibroid embolization: bulk symptoms, pain or heavy menstrual bleeding attributed to fibroids, with imaging confirmation;
* Patient must be able to provide written, informed consent

Exclusion Criteria:

* Documented of allergy or intolerance to lidocaine or other amide-type anesthetics;
* Personal or familial history of malignant familial hyperthermia;
* Documented history of second or third atrio-ventricular heart block
* Contra-indication to uterine fibroid embolization : active infection, suspected malignancy, coagulopathy, pregnancy or desire to preserve fertility, large pedunculated sub-serosal fibroid.
* History of previous uterine fibroid embolization.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Post-Procedural Pain at 4 hours | 4h post-procedure
  Pain will be evaluated using a validated 100mm Visual Analog Scale (VAS) filled by patients at 4h, 7h and 24h post-procedure. At 4h, patients will report the worst pain they experienced since end of procedure. At 7h and 24h, pain at time of assessment will be recorded.
Post-Procedural Pain at 7 hours | 7h post-procedure
  Pain will be evaluated using a validated 100mm Visual Analog Scale (VAS)

SECONDARY OUTCOMES:
Hospital length-of-stay | 24 hours post-intervention
  Estimated in hours, the length-of-stay will be evaluated from the end of procedure to discharge.
Narcotic dose | 24 hours post-intervention
  The total amount on narcotic doses administered to patient during the first 24hours post-procedure will be recorded.
Post-Procedural Pain at 24 hours | 24 hours post-procedure
  Pain will be evaluated using a validated 100mm Visual Analog Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Dheeraj Rajan, MD, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Keyoung JA, Levy EB, Roth AR, Gomez-Jorge J, Chang TC, Spies JB. Intraarterial lidocaine for pain control after uterine artery embolization for leiomyomata. J Vasc Interv Radiol. 2001 Sep;12(9):1065-9. doi: 10.1016/s1051-0443(07)61592-9. PMID 11535769
- [Background] Zhan S, Li Y, Wang G, Han H, Yang Z. Effectiveness of intra-arterial anesthesia for uterine fibroid embolization using dilute lidocaine. Eur Radiol. 2005 Aug;15(8):1752-6. doi: 10.1007/s00330-005-2686-0. Epub 2005 Feb 5. PMID 15696287
- [Background] Baird DD, Dunson DB, Hill MC, Cousins D, Schectman JM. High cumulative incidence of uterine leiomyoma in black and white women: ultrasound evidence. Am J Obstet Gynecol. 2003 Jan;188(1):100-7. doi: 10.1067/mob.2003.99. PMID 12548202
- [Background] Pinto I, Chimeno P, Romo A, Paul L, Haya J, de la Cal MA, Bajo J. Uterine fibroids: uterine artery embolization versus abdominal hysterectomy for treatment--a prospective, randomized, and controlled clinical trial. Radiology. 2003 Feb;226(2):425-31. doi: 10.1148/radiol.2262011716. PMID 12563136
- [Background] Hehenkamp WJ, Volkers NA, Donderwinkel PF, de Blok S, Birnie E, Ankum WM, Reekers JA. Uterine artery embolization versus hysterectomy in the treatment of symptomatic uterine fibroids (EMMY trial): peri- and postprocedural results from a randomized controlled trial. Am J Obstet Gynecol. 2005 Nov;193(5):1618-29. doi: 10.1016/j.ajog.2005.05.017. PMID 16260201
- [Background] Hehenkamp WJ, Volkers NA, Birnie E, Reekers JA, Ankum WM. Symptomatic uterine fibroids: treatment with uterine artery embolization or hysterectomy--results from the randomized clinical Embolisation versus Hysterectomy (EMMY) Trial. Radiology. 2008 Mar;246(3):823-32. doi: 10.1148/radiol.2463070260. Epub 2008 Jan 9. PMID 18187401
- [Background] Volkers NA, Hehenkamp WJ, Birnie E, Ankum WM, Reekers JA. Uterine artery embolization versus hysterectomy in the treatment of symptomatic uterine fibroids: 2 years' outcome from the randomized EMMY trial. Am J Obstet Gynecol. 2007 Jun;196(6):519.e1-11. doi: 10.1016/j.ajog.2007.02.029. PMID 17547877
- [Background] Ananthakrishnan G, Murray L, Ritchie M, Murray G, Bryden F, Lassman S, Lumsden MA, Moss JG. Randomized comparison of uterine artery embolization (UAE) with surgical treatment in patients with symptomatic uterine fibroids (REST trial): subanalysis of 5-year MRI findings. Cardiovasc Intervent Radiol. 2013 Jun;36(3):676-81. doi: 10.1007/s00270-012-0485-y. Epub 2012 Oct 16. PMID 23070101
- [Background] Edwards RD, Moss JG, Lumsden MA, Wu O, Murray LS, Twaddle S, Murray GD; Committee of the Randomized Trial of Embolization versus Surgical Treatment for Fibroids. Uterine-artery embolization versus surgery for symptomatic uterine fibroids. N Engl J Med. 2007 Jan 25;356(4):360-70. doi: 10.1056/NEJMoa062003. PMID 17251532
- [Background] Moss JG, Cooper KG, Khaund A, Murray LS, Murray GD, Wu O, Craig LE, Lumsden MA. Randomised comparison of uterine artery embolisation (UAE) with surgical treatment in patients with symptomatic uterine fibroids (REST trial): 5-year results. BJOG. 2011 Jul;118(8):936-44. doi: 10.1111/j.1471-0528.2011.02952.x. Epub 2011 Apr 12. PMID 21481151
- [Background] Spencer EB, Stratil P, Mizones H. Clinical and periprocedural pain management for uterine artery embolization. Semin Intervent Radiol. 2013 Dec;30(4):354-63. doi: 10.1055/s-0033-1359729. PMID 24436562
- [Background] Pron G, Bennett J, Common A, Wall J, Asch M, Sniderman K; Ontario Uterine Fibroid Embolization Collaboration Group. The Ontario Uterine Fibroid Embolization Trial. Part 2. Uterine fibroid reduction and symptom relief after uterine artery embolization for fibroids. Fertil Steril. 2003 Jan;79(1):120-7. doi: 10.1016/s0015-0282(02)04538-7. PMID 12524074
- [Background] Walker WJ, Pelage JP. Uterine artery embolisation for symptomatic fibroids: clinical results in 400 women with imaging follow up. BJOG. 2002 Nov;109(11):1262-72. doi: 10.1046/j.1471-0528.2002.01449.x. PMID 12452465
- [Background] van der Kooij SM, Moolenaar LM, Ankum WM, Reekers JA, Mol BWJ, Hehenkamp WJK. Epidural analgesia versus patient-controlled analgesia for pain relief in uterine artery embolization for uterine fibroids: a decision analysis. Cardiovasc Intervent Radiol. 2013 Dec;36(6):1514-1520. doi: 10.1007/s00270-013-0607-1. Epub 2013 Apr 11. PMID 23576212
- [Background] Rasuli P, Jolly EE, Hammond I, French GJ, Preston R, Goulet S, Hamilton L, Tabib M. Superior hypogastric nerve block for pain control in outpatient uterine artery embolization. J Vasc Interv Radiol. 2004 Dec;15(12):1423-9. doi: 10.1097/01.RVI.0000137406.09852.A4. PMID 15590800
- [Background] Guthaner DF, Silverman JF, Hayden WG, Wexler L. Intraarterial analgesia in peripheral arteriography. AJR Am J Roentgenol. 1977 May;128(5):737-9. doi: 10.2214/ajr.128.5.737. PMID 404894
- [Background] Widrich WC, Singer RJ, Robbins AH. The use of intra-arterial lidocaine to control pain due to aortofemoral arteriography. Radiology. 1977 Jul;124(1):37-41. doi: 10.1148/124.1.37. PMID 325598
- [Background] Widrich WC, Robbins AH, Goldstein SA, Singer RJ. Adjuvant intra-arterial lidocaine in aortofemoral arteriography: some further observations. Radiology. 1978 Nov;129(2):371-3. doi: 10.1148/129.2.371. PMID 360272
- [Background] Cranston PE. Lidocaine analgesia in peripheral angiography: a confirmation of effectiveness. South Med J. 1982 Oct;75(10):1229-31. doi: 10.1097/00007611-198210000-00018. No abstract available. PMID 7123294
- [Background] Gordon IJ, Westcott JL. Intra-arterial lidocaine: an effective analgesic for peripheral angiography. Radiology. 1977 Jul;124(1):43-5. doi: 10.1148/124.1.43. PMID 866655
- [Background] Molgaard CP, Teitelbaum GP, Pentecost MJ, Finck EJ, Davis SH, Dziubinski JE, Daniels JR. Intraarterial administration of lidocaine for analgesia in hepatic chemoembolization. J Vasc Interv Radiol. 1990 Nov;1(1):81-5. doi: 10.1016/s1051-0443(90)72508-0. PMID 1966862
- [Background] Hartnell GG, Gates J, Stuart K, Underhill J, Brophy DP. Hepatic chemoembolization: effect of intraarterial lidocaine on pain and postprocedure recovery. Cardiovasc Intervent Radiol. 1999 Jul-Aug;22(4):293-7. doi: 10.1007/s002709900391. PMID 10415218
- [Background] Breivik H, Borchgrevink PC, Allen SM, Rosseland LA, Romundstad L, Hals EK, Kvarstein G, Stubhaug A. Assessment of pain. Br J Anaesth. 2008 Jul;101(1):17-24. doi: 10.1093/bja/aen103. Epub 2008 May 16. PMID 18487245
- [Background] Pron G, Mocarski E, Bennett J, Vilos G, Common A, Zaidi M, Sniderman K, Asch M, Kozak R, Simons M, Tran C, Kachura J; Ontario UFE Collaborative Group. Tolerance, hospital stay, and recovery after uterine artery embolization for fibroids: the Ontario Uterine Fibroid Embolization Trial. J Vasc Interv Radiol. 2003 Oct;14(10):1243-50. doi: 10.1097/01.rvi.0000092664.72261.f9. PMID 14551270
- See also: UHN research ethics board contact information — http://www.uhnresearch.ca/reb/rebcontactus.htm